CLINICAL TRIAL: NCT06855095
Title: Absorbed Tumor Dose in Peptide Receptor Radionuclide Therapy with Long-acting Somatostatin Analogues - ATSA Trial
Acronym: ATSA
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Neuroendocrine Tumor Research Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N23PRR
Record Dates: First submitted 2023-10-25; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Neuroendocrine Tumors; Neuroendocrine Tumor Grade 1; Neuroendocrine Tumor Grade 2; Neuroendocrine Neoplasm
Keywords: Peptide Receptor Radionuclide Therapy; PRRT; Lutetium; DOTATATE
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Somatostatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): In this arm, patients without any LA-SSA treatment for at least 3 months prior to PRRT are included.
- 2A - LA-SSA injection 4-6 weeks before PRRT (Active Comparator): In this arm, patients on LA-SSA treatment for at least 3 months prior to PRRT are included and will receive the last LA-SSA injection 4-6 weeks before PRRT.
  Interventions: Drug: Somatostatin analog
- 2B - LA-SSA injection 1-7 days before PRRT (Experimental): In this arm, patients on LA-SSA treatment for at least 3 months prior to PRRT are included and will receive the last LA-SSA injection 4-6 weeks before PRRT.
  Interventions: Drug: Somatostatin analog

INTERVENTIONS:
Drug: Somatostatin analog — Timing of LA-SSA injection prior to PRRT (either 4-6 weeks or 1-7 days).
  Arms: 2A - LA-SSA injection 4-6 weeks before PRRT; 2B - LA-SSA injection 1-7 days before PRRT

SUMMARY:
According to current guidelines, patients have to withhalt long-acting somatostatin analogues (LA-SSA) for 4-6 weeks prior to every 177Lutetium-DOTATATE administration. The primary objective of the study is to investigate the effect of LA-SSA on the absorbed dose in tumor lesions during PRRT.

DETAILED DESCRIPTION:
The study population includes all patients aged over 18 with a neuroendocrine tumor grade I and II and a clinical indication for PRRT. Patients treated for at least three months with LA-SSA are randomized over two interventional arms: one arm where patients discontinue LA-SSA 4-6 weeks before the first PRRT treatment and one arm where patients continue LA-SSA treatment and receive the first PRRT administration within one week after the most recent LA-SSA injection. Patients in the control arm who have not been treated with LA-SSA in the last three months will start PRRT according to standard local protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Able to provide spoken and written informed consent for the trial;
* Histopathological confirmed neuroendocrine tumor;
* Fulfill the clinical criteria for PRRT;
* At least one soft tissue lesion > 2 cm;
* Aimed administered activity of 7400 MBq;
* ECOG score (performance status) 0-2.

Exclusion Criteria:

* Not possible to discontinue LA-SSA for 4-6 weeks;
* Use of short-acting SSAs;
* Pregnancy and lactating female patients;
* Inability to comply to the study procedures;
* Factors that might affect the biodistribution (for example, indication for furosemide directly after PRRT infusion, limited fluid intake, any renal catheters, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Effect of continued LA-SSA use on the absorbed dose in tumor lesions during PRRT. | SPECT/CT after 4h, 24h, and 5-7 days post-injection

SECONDARY OUTCOMES:
Effect of continued LA-SSA use on the absorbed dose in normal tissues during PRRT. | SPECT/CT after 4h, 24h, and 5-7 days post-injection and blood samples at 2h, 4h, 24h and 5-7 days post-injection
Effect of continued LA-SSA use on the tumor-to-background ratio. | SPECT/CT after 4h, 24h, and 5-7 days post-injection
Effect of continued LA-SSA use on population pharmacokinetic parameters of [177Lu]Lu-HA-DOTATATE. | Blood samples at 2h, 4h, 24h and 5-7 days post-injection

OTHER OUTCOMES:
HRQoL assessments | At baseline, on the day of PRRT administration, 3 weeks after PRRT

CONTACTS AND LOCATIONS:
Locations (1):
- Antoni van Leeuwenhoek, Amsterdam, Netherlands